CLINICAL TRIAL: NCT06528704
Title: The Impact of Real Time Ventilation Feedback on Ventilation Rate and Tidal Volume During Cardiac Arrest.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONZ-2023-0613
Record Dates: First submitted 2024-05-22; First posted 2024-07-30 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ventilation feedback (Experimental): First, ventilation without feedback, hereafter ventilation with feedback
  Interventions: Device: Ventilation feedback device

INTERVENTIONS:
Device: Ventilation feedback device — Device showing delivered ventilation frequency and volume.

SUMMARY:
During out-of-hospital cardiopulmonary resuscitation, patient are first ventilated without ventilation feedback (but with a flowsensor connected), hereafter patients are ventilated with the use of ventilation feedback.

DETAILED DESCRIPTION:
During cardiac arrest, patients are intubated, ventilation is performed using a manual resuscitator. Hereafeter, a flowsensor is connected. During the first cycle, patients are ventilated without any feedback (whilst the sensor is recording the delivered ventilation). During the second cycle, realtime delivered flow is shown on the screen, informing the user on the delivered ventilation volume and ventilation rate. Data is saved automatically after use.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

Traumatic cardiac arrest Inability to intubate patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Delivered ventilation frequency | 2 minutes
  Measured ventilation frequency (with or without ventilation feedback)
Delivered ventilation volume | 2 minutes
  Measured ventilation volume (with or without ventilation feedback)

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - AZ Zeno, Knokke, West-Vlaanderen
  - Ghent University Hospital, Ghent

IPD SHARING:
Plan to Share IPD: No